CLINICAL TRIAL: NCT06723535
Title: An Open-Label, Single-Dose, Phase 1 Study to Evaluate the Pharmacokinetics and Safety of BMS-986278 in Participants With Normal Renal Function, Participants With Severe Renal Impairment, and Participants With End-Stage Renal Disease on Intermittent Hemodialysis
Brief Title: A Study to Evaluate BMS-986278 in Participants With Normal Renal Function, Severe Renal Impairment, or End-Stage Renal Disease on Intermittent Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM027-1014
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Kidney Failure, Chronic; Healthy Volunteers; Renal Impairment
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A and C (Experimental)
  Interventions: Drug: BMS-986278
- Group B: Period 1 (Experimental)
  Interventions: Drug: BMS-986278
- Group B: Period 2 (Experimental)
  Interventions: Drug: BMS-986278

INTERVENTIONS:
Drug: BMS-986278 — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess the effect of severe renal impairment (RI) and end-stage renal disease (ESRD) with intermittent hemodialysis (IHD) on the pharmacokinetics and safety of BMS-986278. This study plans to use a staged design based on RI severity.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 45 kg/m2 inclusive, and body weight ≥ 50 kg at screening. Note: for ESRD participants, this body weight should be the prescription dry weight.
* Severe Renal Impaired Participants:

  1. Participant has a supine SBP ≥ 90 and ≤ 180 mmHg, supine DBP ≥ 60 and ≤ 100 mmHg, and heart rate ≥ 40 and ≤ 110 beats per minute.
  2. Participant has severe RI as defined by an eGFR ˂ 30 mL/min and not requiring dialysis at screening.
  3. Participant must be medically stable for at least 1 month before study intervention administration.
* Participants with ESRD:

  1. Participant has ESRD as defined by an eGFR < 15 mL/min at screening.
  2. Participant required to be on intermittent hemodialysis, an average of 3 hemodialysis treatments per week prior to screening.
  3. Participant has demonstrated adequate hemodialysis measurements (at least 2 Kt/V measurements ≥ 1.2 or 2 urea reduction ratio measurements ≥ 65%) within the 3 months prior to screening.
* Healthy participant should have a supine SBP ≥ 90 and ≤ 160 mm Hg, supine DBP ≥ 50 and ≤ 100 mm Hg, and heart rate ≥ 40 and ≤ 100 beats per minute.
* Healthy participants should have normal renal function, as defined by having an eGFR ≥ 90 mL/min eGFR at screening (calculated using the CKD-EPI equation).

Exclusion Criteria:

* Participant with any significant medical condition, laboratory abnormality, or psychiatric illness.
* Any surgical or medical condition(s) possibly affecting drug absorption, distribution, metabolism, or excretion (eg, bariatric procedure or cholecystectomy).
* Individuals who are of childbearing potential, breastfeeding, or currently pregnant.
* Other protocol defined inclusion/exclusion criteria apply.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-12-07 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to Day 8
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] | Up to Day 8
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] | Up to Day 8

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 28 days following discontinuation of dosing
Number of participants with physical examination abnormalities | Up to Day 8
Number of participants with vital sign abnormalities | Up to Day 8
Number of participants with 12-lead electrocardiogram (ECG) abnormalities | Up to Day 8
Number of participants with clinical laboratory abnormalities | Up to Day 8
Time of maximum observed concentration (Tmax) | Up to Day 8
Terminal elimination half-life (T-HALF) | Up to Day 8
Apparent body clearance (CLT/F) | Up to Day 8
Apparent volume of distribution of terminal phase (Vz/F) | Up to Day 8
Concentration of BMS-986278 in dialysate | Up to Day 8
Total amount recovered in dialysate (DR) | Up to Day 8
Total percent of administered dose recovered in dialysate (%DR) | Up to Day 8
Free fraction of unbound drug (Fu) | Up to Day 8
Unbound Cmax (Cmax_u) | Up to Day 8
Unbound AUC(0-T) (AUC(0-T) _u) | Up to Day 8
Unbound AUC(INF) (AUC(INF)_u) | Up to Day 8
Unbound CLT/F (CLT/F_u) | Up to Day 8
Unbound Vz/F (Vz/F_u) | Up to Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - Local Institution - 0002, Miami, Florida
  - Local Institution - 0003, Miami, Florida
  - Local Institution - 0004, Orlando, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com